CLINICAL TRIAL: NCT03795051
Title: Precise Coil Positioning in Navigated Transcranial Magnetic Stimulation (nTMS) in Medication- Resistant Major Depressive Disorder (MDD): A Feasibility Study
Brief Title: Coil Positioning in Navigated Transcranial Magnetic Stimulation Feasibility in Depression Patients Trial
Acronym: CONFIDENT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Magstim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MGS-2018-SS
Record Dates: First submitted 2018-11-14; First posted 2019-01-07 (Actual); Last update posted 2020-01-03 (Actual); Status verified 2020-01

CONDITIONS: Depressive Disorder, Major
Keywords: Transcranial Magnetic Stimulation; Navigated Transcranial Magnetic Stimulation
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Navigated TMS (Experimental): Each participant will receive 30 sessions of 10 Hz or 20 Hz navigated transcranial magnetic stimulation over the left DLPFC.
  Interventions: Device: Navigated Transcranial Magnetic Stimulation

INTERVENTIONS:
Device: Navigated Transcranial Magnetic Stimulation — This study is a feasibility trial. Each participant will receive 30sessions of 10 Hz or 20 Hz rTMS over the left DLPFC. The rTMS interventions will be guided by a neuronavigation system (StimGuide TMS Navigation System, Magstim, Ltd. Carmarthenshire, UK) for navigation to the treatment location and to ensure consistent placement and orientation of the coil during and between each session. For the purpose of this protocol, these sessions are referred to as nTMS.

SUMMARY:
The objective of this study is to evaluate the feasibility of adding a navigational system to traditional repetitive Transcranial Magnetic Stimulation (rTMS, referred to in this application as nTMS) as a way to establish and maintain precise coil positioning (contact, rotation, and tilt) and consistent brain region targeting throughout a nTMS treatment session and in subsequent nTMS sessions.

DETAILED DESCRIPTION:
Objective: The objective of this study is to evaluate the feasibility of adding a navigational system to traditional repetitive Transcranial Magnetic Stimulation (rTMS, referred to in this application as nTMS) as a way to establish and maintain precise coil positioning (contact, rotation, and tilt) and consistent brain region targeting throughout a nTMS treatment session and in subsequent nTMS sessions. Success will be evaluated via data analysis of information captured during nTMS, which will evaluate coordinates, contact, rotation, and tilt parameters of the stimulation pulses delivered. The study will be conducted with patients who have been selected as traditional rTMS candidates and have met the criteria for rTMS, which includes, but is not limited to the following: Adults with Major Depressive Disorder (MDD) who have failed to achieve satisfactory improvement from prior antidepressant medication in the current episode. For the purposes of this study, nTMS is referring to the use of a navigation device in combination with delivery of traditional rTMS.

Aim 1: Determine the percentage of successful nTMS treatment sessions. A successful nTMS treatment session is defined as the following: 80% of the TMS pulse trains are delivered while the coil is within acceptance criteria measured by tracking the following parameters: coil deviations from digitally saved target location, which includes contact (mm), rotation (°), and tilt (°) parameters. The acceptance criteria are met with coil position at the time of pulse delivery as follows: coil rotation within ±15° of target; coil tilt within ±15° of target; in-plane deviation within ±5mm of target; contact deviation within ±2mm of target.

Aim 2: Determine Patient Health Questionnaire (PHQ-9) change measured weekly from baseline to after 30 sessions of nTMS, collect Patient comfort data, measure Operator confidence and collect coil position data for nTMS sessions to determine future product improvements and clinical studies.

The goal of this proposal is to establish nTMS as a means of precise administration of transcranial magnetic stimulation. Ultimately, data from this study will be used to design larger, comparative studies to establish superior efficacy profiles in the treatment of MDD.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of medication-resistant MDD,
* Age 18 years or older
* Normal findings in the medical history, physical, and neurological examination

Exclusion Criteria:

* History of seizure disorder
* History of neuroleptic medications/prior use of neuroleptics
* Presence of implanted medical pump, metal plate, or metal object in skull or eye
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-09 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Percentage of successful nTMS treatment sessions | The number of successful treatment sessions will be assessed after 6 weeks of treatment. Only data from week 2 through 6 will be included (approximately 25 treatment sessions). (Example 20 out of 25 sessions were successful.)
  The primary outcome measure will be the percentage of successful nTMS treatment sessions pooled from sessions 6 through 30 for each study subject. A successful nTMS treatment session is defined as: 80% of the TMS pulse trains are delivered while the coil is within acceptance criteria measured by tracking the following parameters: coil deviations from digitally saved target location, which includes contact (mm), rotation (°), and tilt (°) parameters. The acceptance criteria are met with coil position at the time of pulse delivery as follows: coil rotation within ±15° of target; coil tilt within ±15° of target; in-plane deviation within ±5mm of target; contact deviation within ±2mm of target.

SECONDARY OUTCOMES:
Operator Confidence | Aproximately 5 months after first patient treatment. After last study patient at site has completed the treatment or has exited the study (expected for May 2019).
  Operator confidence will be measured on a scale of 1 to 5; 1 being not confident at all in using StimGuide to consistently find the treatment site and deliver therapy to 5 being very confident in using StimGuide to consistently find the treatment site and deliver therapy.
Patient Comfort | After last treatment has been completed; approximately six week after treatment start
  Patient comfort measured on a scale from 1 to 5; with 1 being uncomfortable and 5 being extremely comfortable
Patient Health Questionnaire 9 (PHQ-9) - Patient Depression Questionnaire | At baseline and after six weeks of treatment
  Patient Health Questionnaire (PHQ-9) change from baseline. The PHQ-9 Patient Depression Questionnaire has 9 questions with a scale range for each question of 0 to 3 (0 = not at all, 1 = several days, 2 = more than half the days, 3 = nearly every day. The maximum summed score (severely depressed) is 27.
Coil Position deviation from target | Coil position deviation: every treatment session during week 2 through 6
  Coil deviation for every pulse train for each patient's nTMS session. Coil deviations from digitally saved target location, which includes contact (mm), rotation (°), and tilt (°) parameters will be measured and reported.

CONTACTS AND LOCATIONS:
Overall Officials: Lothar Krinke, PhD, Principal Investigator — Magstim
Locations (2):
- United States (2):
  - Georgia Behavioral Health Professionals, Atlanta, Georgia
  - Georgia Behavioral Health Professionals, Dunwoody, Georgia

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/51/NCT03795051/Prot_ICF_000.pdf